CLINICAL TRIAL: NCT00348322
Title: An Evaluation of the Safety and Efficacy of Systane Free FID 105783 - II
Brief Title: Safety/Efficacy of Systane Free vs Refresh Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-06-22
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Systane Free Lubricant Eye Drops

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Systane Free FID 105783 in comparison to Refresh Tears Lubricant Eye Drops (Allergan) in a specified population of dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* > = 3 stain using NEI grid and need artificial tears at least some of the time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Corneal Staining change from baseline

SECONDARY OUTCOMES:
Comfort, Conjunctival Staining

CONTACTS AND LOCATIONS:
Overall Officials: Mike Christensen, Study Director — Alcon Research
Locations (1):
- El Paso Facility, El Paso, Texas, United States